CLINICAL TRIAL: NCT00004696
Title: Study of Morphine in Postoperative Infants to Allow Normal Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized
Other Study IDs: 199/13359; CHMC-S-FDR001015; CHMC-S-IRB-022-9801; CHMC-S-IRB-148-9706
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-05

CONDITIONS: Infant, Newborn, Diseases; Pain
Keywords: disease-related problem/condition; pain; intraoperative/postoperative complications; rare disease
MeSH Terms: conditions — Infant, Newborn, Diseases; Pain; Postoperative Complications; Rare Diseases | interventions — Morphine

INTERVENTIONS:
Drug: morphine

SUMMARY:
OBJECTIVES: I. Compare nonmechanically ventilated infants who receive morphine postoperatively as intermittent intravenous bolus doses or as a continuous intravenous infusion targeted to reach a steady-state concentration.

II. Assess ventilation (blood gases, continuous oximetry, and CO2 response curves) and analgesia (infant pain score) between the two treatment groups of infants.

III. Compare ventilation parameters (blood gases, CO2 response curves, and time to wean from assisted mechanical ventilation) in cyanotic and acyanotic infants after thoracotomies.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a two part study. Infants are stratified by age (1-30 days vs 31-180 days vs 181-365 days) and by type of surgery. Infants are randomly assigned to one of two treatment arms.

In part I, following major thoracic, abdominal, or cardiac surgery, infants are randomized to receive either continuous IV morphine infusions (arm I) or to receive morphine by single IV bolus doses every 2-3 hours (arm II).

In part II, cyanotic and acyanotic infants following thoracotomy receive morphine by 2 loading doses over 15 minutes and then by continuous IV infusion.

Patients are followed for at least 2 days.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Infants scheduled for surgery with postoperative inpatient care
* Must be born after 35 weeks or more gestational age
* No prenatal opiate exposure

Part I patients:

* Less than 12 months of age undergoing surgeries involving major thoracic, abdominal, or cardiac procedures
* No pneumonectomy, tracheal or bronchial stenosis reconstruction, diaphragmatic hernia repair, or surgeries resulting in high intraabdominal pressure (closure of large gastroschisis or omphalocele defects)
* No hepatic or renal transplantation

Part II patients:

* Less than 3 months of age undergoing surgeries using a thoracotomy approach
* Cyanotic congenital heart disease having palliative systemic to pulmonary artery shunts created OR Thoracotomy for repair of acyanotic lesions (e.g., repairs of coarctation of the aorta, tracheoesophageal fistula repair, PDA ligation)

--Patient Characteristics--

* Age: Part I: Less than 12 months Part II: Less than 3 months
* Hepatic: Normal hepatic function tests
* Renal: Normal renal function tests
* Pulmonary: No pulmonary disease causing baseline hypercarbia
* No pulmonary hypertension contraindicating use of 5% CO2 in rebreathing studies

Other:

* No allergy to morphine
* No severe developmental delay that precludes analgesia scoring

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 1994-08; Study Completion 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Anne M. Lynn, Study Chair — Seattle Children's Hospital

REFERENCES:
- [Background] Lynn A, Nespeca MK, Bratton SL, Strauss SG, Shen DD. Clearance of morphine in postoperative infants during intravenous infusion: the influence of age and surgery. Anesth Analg. 1998 May;86(5):958-63. doi: 10.1097/00000539-199805000-00008. PMID 9585276